CLINICAL TRIAL: NCT00436423
Title: A Phase Ⅱ Study of Gemcitabine Combination With TS-1 in Patient With Advanced or Recurred Pancreatic Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Korea University Anam Hospital (Other)
Collaborators: Seoul National University Hospital (Other); Seoul Municipal Boramae Hospital (Unknown); Konkuk University Hospital (Other); Korea University Ansan Hospital (Other); Seoul National University Bundang Hospital (Other); Korea University Guro Hospital (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AN0561-008
Record Dates: First submitted 2007-02-16; First posted 2007-02-19 (Estimated); Last update posted 2007-11-01 (Estimated); Status verified 2007-10

CONDITIONS: Pancreatic Neoplasm; Neoplasm Metastasis
Keywords: pancreatic neoplasm; drug therapy; gemcitabine; TS-1
MeSH Terms: conditions — Pancreatic Neoplasms; Neoplasm Metastasis | interventions — Gemcitabine; titanium silicide

ARMS (1):
- 1 (Experimental): Gemcitabine with TS-1
  Interventions: Drug: gemcitabine, TS-1

INTERVENTIONS:
Drug: gemcitabine, TS-1

SUMMARY:
The primary objective of the study is to Evaluate the response rate of Gemcitabine with TS-1 in Korean patient with advanced but inoperable, metastatic or recurrent pancreatic cancer who is not receiving anti cancer therapy.

DETAILED DESCRIPTION:
To date, curative treatment of pancreatic cancer is surgery.But patients with operable indication are rare, most of patients present with locally advanced or general advanced stage at diagnosis. Thus the majority of patients need chemotherapy.But efficacy outcomes have not seemed to increase overall survival comparing with none treated control group.In Korea the incidence of pancreatic cancer increases steadily. Prognosis is poor. So now the effective treatment is necessary.There are no phase 2 trialsabout combining gemcitabine and TS-1 against advanced pancreatic cancer.according to phase 1 trial of advanced pancreatic cancer (nakamura et al)toxicities more than 3 grade are neutropenia, anemia, thrombocytopenia, anorexia, etc that can be treated.Phase 1 trial is not study to evaluate the response rate. But among 21 patients who can be evaluated the response rate, 10 patients have Partial response or Complete response.This combination therapy seemed to havetolerable toxicity and remarkable therapeutic effect for locally advanced or metastatic pancreatic cancer.So therapy combining gemcitabine with TS-1 is expected synergic and additional effect.

This trial is phase 2, open-label, multi-center, single arm study The total sample size will be 38 patients. Patient will be administered chemotherapy until disease progression. Gemcitabine will be administered at a dose of 1000 mg/m2 every 3weeks (on day 1 of each cycle) TS-1 will be administered 80 mg/m2 orally twice daily for 14 days every 3 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. histologically or cytologically confirmed adenocarcinoma with inoperable locally advanced or metastatic or recurrent pancreatic cancer after previous operation or radiation therapy
2. performance statues 0,1 or 2 on the ECOG scale
3. life expectance of at least 3 months
4. adequate organ function including the following <adequatebone marrow function> Absolute neutrophil count(ANC) ≥ 1.5 � 109/L Platelets ≥ 100 � 109/L Hemoglobin ≥ 9 g/dL <adequate hepatic function> Serum AST, ALT< 5 X upper limit of normal(ULT) serum bilirubin< 2 X ULT Patient with obstructive jaundice and serum bilirubin more than double of upper limit of normal have to drain bile internally or externally before enrolment.

   <adequate renal function> Creatinine < 1.5 X ULT
5. consent form which is voluntarily signed by patients or legal representative
6. men or women , age 18
7. previous chemotherapy is not allowed. But previous adjuvant or neo adjuvant chemotherapy is allowed Patient must completed previous adjuvant or neo adjuvant chemotherapy at least one month.

   Patient must have recovered from the toxic effect of the treatment But patient who are to receive gemcitabin and TS-1 on previous adjuvant or neo adjuvant chemotherapy must not be enrolled.
8. Measurable disease, according to the response Evaluation criteria in solid tumors(RECIST), assessed using imaging techniques(CT or MRI)

Exclusion Criteria:

1. have received treatment within the last 30 days of study enrolment with a drug that has not received approval for any indication
2. heart failure, angina pectoris or arrhythmia which is uncontrolledwith medication within the previous 6 month .
3. serious neurological or mental disorder.
4. active infection that would compromise the patient's ability to stand the study, at the discretion of the investigator.
5. uncontrolled diabetes.
6. serious concomitant disorders that would compromisethe safety of the patient or compromise the patient's ability to complete the study, at the discretion of the investigator.
7. pregnancy
8. breast feeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2006-03

PRIMARY OUTCOMES:
Response rate by RECIST criteria

SECONDARY OUTCOMES:
Describe quantitative and qualitative toxicity of gemcitabine with TS-1
Evaluate the following efficacy measure Duration of response,Time to treatment failure,Time to documented disease progression, Overall survival

CONTACTS AND LOCATIONS:
Overall Officials: YeulHong Kim, professor, Principal Investigator — Korea University Anam Hospital
Locations (1):
- YeulHong Kim, Seoul, South Korea